CLINICAL TRIAL: NCT07290790
Title: A Prospective, Multicenter, Randomized, Post-market Clinical Investigation to Assess the Accuracy of Different Tooth Movements for Patients Undergoing Clear Aligner Therapy (CAT) With SureSmile® Clear Aligners With Three Different Trimlines.
Brief Title: A Prospective Multicenter Clinical Investigation Evaluating the Accuracy of the Trimline Design When Treated With SureSmile® Aligners.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-OR-25-002
Record Dates: First submitted 2025-12-15; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Scalloped trimline design (Experimental): SureSmile® Clear Aligner (Group 1) with scalloped trimline design
  Interventions: Device: SureSmile® Clear Aligners
- Straight trimline design (Experimental): SureSmile® Clear Aligner (Group 2) with straight trimline design
  Interventions: Device: SureSmile® Clear Aligners
- Extended trimline design (Experimental): SureSmile® Clear Aligner (Group 3) with extended trimline design (2 mm)
  Interventions: Device: SureSmile® Clear Aligners

INTERVENTIONS:
Device: SureSmile® Clear Aligners — SureSmile® Clear Aligners are Custom-made (EU)/patient matched (US) medical devices made to fit appliance with different diameters and lengths to accommodate subjects with different mouth shapes and sizes.
  This clinical investigation consists of three different trimline designs groups:
  * SureSmile aligner Scallop trimline design
  * SureSmile aligner Straight trimline design
  * SureSmile aligner Straight extended trimline design
  All pre-treatment, treatment, and post-treatment protocols and materials used in all groups are identical, except for the type of trimline design.

SUMMARY:
This is a three-armed, multicenter clinical study evaluating the SureSmile clear aligner medical device. The primary objective is to confirm the safety and assess the accuracy of different tooth movements. In addition, the study will investigate and compare three different trimline designs: Scalloped, Straight, and Straight Extended.

ELIGIBILITY:
Inclusion Criteria:

* Subject willing to participate in the clinical investigation, able to understand the intent risks and benefits of the clinical investigation as well as associated time commitment and follow-ups visits.
* Subject has signed and dated the informed consent form (ICF) .
* Subject aged 18 years or above at time of informed consent.
* Subject has permanent dentition (i.e., all 2nd molars).
* Subject with a dental malocclusion, consistent with Levels 1 and 2 case complexity and within the clinical references as defined in the SureSmile Case Selection Guide.

  * Crowding or spacing must be ≤6mm present in one or both arches consistent with level 1 and 2 of case complexity.
  * Midline deviation must be ≤3 mm consistent with level 1 and 2 of case complexity.
  * Overjet must be ≤4 mm consistent with level 1 and 2 case complexity.
  * Overbite must be ≤3 mm consistent with level 1 and 2 case complexity.
  * Anterior open bite must be ≤1 mm, consistent with level 1 and 2 case complexity.
* Intermaxillary elastics may be included within the treatment plan to support sagittal, vertical, or transverse correction within the limits defined under exclusion criteria.

Exclusion Criteria:

* Subjects unlikely to comply with investigational procedures, or unlikely to come back for follow-up visits, as judged by the Investigator.
* Subject that presents a dental malocclusion classified as level 3 case complexity, as defined in the SureSmile Case Selection Guide.
* Subjects who have completed aligner therapy within the last 12 months or who are in active orthodontic treatment.
* Subjects with active periodontal disease or other unresolved dental conditions such as active cavities, active periodontal disease.
* Subjects with treatment plans requiring transverse correction requiring expansion greater than 4 mm per arch or 2 mm per quadrant, or any skeletal transverse correction.
* Treatment plans requiring sagittal correction exceeding a half-cusp discrepancy (i.e., >½ unit) in molar or canine relationships.
* Subjects with treatment plans require vertical correction beyond Level 1 and 2 thresholds (i.e., overbite >3 mm or anterior/posterior open bite >1 mm), or vertical elastics exceeding 3 mm.
* TMJ (Temporo-Mandibular Join) disorders or history of headaches or migraines.
* Participants with known history of plastic allergies.
* Subjects with presence of skeletal discrepancies necessitating orthognathic surgery, rapid palatal expansion, other orthopedic intervention, unilateral or bilateral cross-bites, mandibular deviations in association with the diagnosed malocclusion
* The use of TADs (Temporary Anchor Devices), plates, other fixed anchorage ancillaries or the use of functional appliances (distalizers, growth modification devices), any approach involving orthopedic or skeletal sagittal correction or the use of hybrid fixed appliances are not considered part of the scope of this clinical investigation and these subjects are not eligible.
* Uncontrolled para-functional habits, e.g., bruxism.
* Any other condition that would make the subject unsuitable for participation, including but not limited to:

  * Unstable psychiatric illness.
  * Recent myocardial infarction (< 3 months*).
  * Recent cerebrovascular accident (< 3 months*).
  * Recent cardiac-valvular prosthesis placement (< 3 months*).
  * Hemorrhagic diathesis.
  * Severe liver dysfunction.
  * Known or suspected current malignancy.
* Known pregnancy at the time of enrolment.
* Previous enrolment in the present clinical investigation.
* Involvement in the planning and conduct of the clinical investigation (applies to both Dentsply Sirona personnel and the clinical investigation site).
* Participation in another clinical investigation that may interfere with the present clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Tooth movement accuracy at subject level across different movement types | At start of aligner treatment and at end of aligner treatment according to predetermined treatment plan (end of aligner treatment is on average 6-18 months after aligner treatment start).
  The primary objective of this clinical investigation is to provide a detailed assessment of tooth movement accuracy at subject level across different movement types. For each patient, all teeth will be evaluated in five dimensions of movement:
  1. Mesiodistal translation [mm]
  2. Buccolingual translation [mm]
  3. Intrusive/extrusive movement [mm]
  4. Mesiodistal angulation [degrees]
  5. Buccolingual torque [degrees]
  Accuracy will be determined by comparing the predicted versus achieved tooth positions for 16 teeth in each subject using the formula:
  "Percentage of accuracy" =100 - [(|predicted-achieved| / |predicted|) *100]" Subject effectiveness is the overall mean of all the collected "Percentage of accuracy" values.

SECONDARY OUTCOMES:
Perceived comfort/pain | Every 8 weeks from start of aligner treatment up to to end of aligner treatment according to predetermined treatment plan (on average 6-18 months). Plus every 8 weeks during refinement period, on average 8-12 weeks.
  Perceived comfort/pain experienced by subjects will be assessed using a Visual Analogue Scale (VAS) with a Wong Baker face.
SureSmile Clear Aligner Refinement rates. | At end of aligner treatment according to predetermined treatment plan (end of aligner treatment is on average 6-18 months after aligner treatment start).
  SureSmile Clear Aligner Refinement rates aim to measure the number of refinements required among three different trimline groups.
Occurrence of Adverse Events, Adverse Device Effects, and Device Deficiencies during the clinical investigation. | From Day 0 up to Retainer Delivery Visit, on average 18 months post Day 0.
  Adverse Events, Adverse Device Effects, and Device Deficiencies spontaneously reported, and collection at each clinical investigation visit.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Costanzo Orthodontics, Fresno, California
  - Center for Orthodontic Excellence, Princeton Junction, New Jersey
  - Brush 365 Dental, Frisco, Texas
- Clinica dental Francesc Batlle, Barcelona, Spain
- The Sanford, Bexleyheath, United Kingdom

IPD SHARING:
Plan to Share IPD: No